CLINICAL TRIAL: NCT04555603
Title: Retrospective Analysis of Axitinib Treatment Optimization and Management of Selected Immune Related Adverse Events of Checkpoints Inhibitors
Brief Title: Axitinib Therapy Management Study
Status: Withdrawn | Type: Observational
Why Stopped: Failed at data quality assurance process before any analyses would be performed
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061096
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; avelumab; pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Inlyta — axitinib
  Other Names: Axitinib as prescribed in the real world
Drug: Bavencio — avelumab
  Other Names: Avelumab as prescribed in the real world
Drug: Keytruda — Pembrolizumab
  Other Names: Pembrolizumab as prescribed in the real world

SUMMARY:
The objectives of the study is to describe axitinib therapy management through use of the data to be generated by ConcertAI

DETAILED DESCRIPTION:
not mandatory

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of aRCC (Stage III, Stage IV (M0) or Stage IV (M1)) at any point
* Age 18 years or older at the time of aRCC diagnosis
* Received a qualifying IO-containing combination (nivolumab and ipilimumab, axitinib and pembrolizumab, or axitinib and avelumab) in the first regimen after aRCC diagnosis or axitinib monotherapy in any line

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: academic and community centers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
To describe type of immune related adverse events and adverse events related to axitinib | during treatment period
  describe type of immune related adverse events and adverse events related to axitinib
To describe the percentage of patients with documentation of dose modifications | during treatment period
  describe dose modifications
To describe the percentage of patients with usage of concomitant high-dose corticosteroid | during treatment period
  descriptive assessment
To describe the percentage of patients alive at pre-specified time points (6 months, 12 months, 18 months, 24 months) from start of the index therapy | during study period
  calculation of overall survival time
To estimate the best overall response (partial response, complete response, progressive disease, or stable disease | during treatment period
  description of overall response
To estimate time to treatment discontinuation | during treatment period
  calculation of duration of treatment
To estimate PFS | during treatment period
  calculation of progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061096